CLINICAL TRIAL: NCT02502786
Title: A Phase II Study of Humanized Monoclonal Antibody 3F8 (Hu3F8) With Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) in the Treatment of Recurrent Osteosarcoma
Brief Title: Humanized Monoclonal Antibody 3F8 (Hu3F8) With Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) in the Treatment of Recurrent Osteosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Children's Hospital Los Angeles (Other); M.D. Anderson Cancer Center (Other); Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-096
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Osteosarcoma
Keywords: Humanized Monoclonal Antibody 3F8 (Hu3F8); Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF); 15-096
MeSH Terms: conditions — Osteosarcoma | interventions — humanized 3F8 anti-GD2 monoclonal antibody; naxitamab; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (1):
- humanized anti-GD2 antibody, hu3F8, when combined with GM-CSF (Experimental): One cycle consists of treatment with hu3F8 at a dose of 2.4mg/kg/dose for 3 days (day 1, 3, and 5) in the presence of subcutaneous (sc) GM-CSF (day -4 through 5). These 3 doses of hu3F8 and 10 days of GM-CSF constitute a treatment cycle. Cycles are repeated at ~2-4 week intervals between first days of hu3F8, through 5 cycles. A maximum of 5 cycles will be administered on protocol. If elevations of amylase and/or lipase (>Grade 1) or clinical signs suggestive of pancreatitis (e.g. upper abdominal pain) occurs, naxitamab and GM-CSF doses should be held until improvement of toxicity to ≤Grade 1 if laboratory elevations and/or pancreatitis is possibly related to either naxitamab or GM-CSF.
  Interventions: Biological: humanized anti-GD2 antibody; Drug: GM-CSF

INTERVENTIONS:
Biological: humanized anti-GD2 antibody
  Other Names: hu3F8
Drug: GM-CSF

SUMMARY:
The purpose of this study is to find out what effect an antibody called Humanized 3F8 (Hu3F8) and a drug called GM-CSF have on the patient and whether it can keep the patient in remission longer and/or prevent recurrence of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent OS. OS must be verified by histopathology review by the site's Department of Pathology. (Patients registered at MSK must have pathology confirmed by MSK Department of Pathology.)
* Patients must be in a ≥2nd complete remission as indicated by appropriate radiologic evaluations at the time of study entry.
* Patients must be ≥ 1 year of age and ≤ to 40 years of age at the time of enrollment.
* Prior therapy: ≥3 weeks should have elapsed since last cytotoxic therapy, immunotherapy or radiation therapy. More than one week should have elapsed since major surgery.

NOTE: Minor surgery (e.g. minor biopsy, central venous catheter placement, shunt revision) is permitted within 1 week prior to enrollment)

* Adequate hematopoietic function defined as:

  * Absolute neutrophil count ≥ 500/ul
  * Absolute lymphocyte count ≥ 500/ul
  * Platelet count ≥ 50,000/ul (transfusion independent)
* Adequate hepatic function as defined by:

  * Total bilirubin of ≤ 1.5 times upper limit of normal (exception is made for patients with Gilbert's syndrome who may be considered eligible if total bilirubin is ≤ 3 times upper limit of normal).
  * AST (SGOT) of ≤ 3 times upper limit of normal
  * ALT (SGPT) of ≤ 3 times upper limit of normal
* Adequate renal function as defined by a serum creatinine of ≤ 1.5 times upper limit of normal
* Adequate cardiac function as defined by a shortening fraction of ≥ 28% or an ejection fraction ≥ 50%
* Adequate pulmonary function as defined by no evidence of dyspnea at rest at no history of exercise intolerance
* Adequate performance status as defined by ECOG score of ≤ 2 or Karnofsky/Lansky score ≥ 50%
* Prior treatment with other anti-GD2 antibodies is allowed (prior treatment with Hu3F8 is NOT allowed), but HAHA antibody titer must be negative
* Women of child-bearing potential must be willing to practice an effective method of birth control while on treatment
* Signed informed consent indicating awareness of the investigational nature of this program

Exclusion Criteria:

* Patients with OS in first complete remission.
* Presence of overt metastatic disease at any site.
* Active life-threatening infection.
* Pregnant women or women who are breast-feeding.
* Inability to comply with protocol requirements.

Ages: 13 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2015-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
event free survival (EFS) | 12 months
  EFS is defined as the time from surgery to relapse or death from any cause, recurrence of tumor or second malignancy.

SECONDARY OUTCOMES:
time to recurrence | 12 months
  Time to recurrence will be estimated using Kaplan-Meier methods. Very few patients are expected to die without relapse (<5%). Recurrence is defined as the radiographic presence of any new lesion that is not attributable to differences in scanning techniques, change in imaging modality or findings thought to represent something other than osteosarcoma, or if a biopsy is performed which shows osteosarcoma.

CONTACTS AND LOCATIONS:
Overall Officials: Filemon Dela Cruz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Children's Hospital of Los Angeles (Data Collection Only), Los Angeles, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD ANDERSON CANCER CENTER (Data Collection Only), Houston, Texas

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/